CLINICAL TRIAL: NCT00391196
Title: A 1-Year, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study To Evaluate The Efficacy And Safety Of CP-945,598 In The Treatment Of Overweight, Oral Agent-Treated Subjects With Type 2 Diabetes Mellitus
Brief Title: A 1-Year Study On The Effects Of CP-945,598 For The Treatment Of Obesity In Overweight Type 2 Diabetic Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5351022
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CP-945,598 (Experimental)
  Interventions: Drug: CP-945,598
- CP-945,598 Treatment B (Experimental): Subjects receive CP-945,598 plus non-pharmacological weight loss program.
  Interventions: Drug: CP-945,598 Treatment B

INTERVENTIONS:
Drug: Placebo — Subjects receive placebo plus non-pharmacological weight loss program.
  Arms: Placebo
Drug: CP-945,598 — Subjects receive CP-945,598 plus non-pharmacological weight loss program.
  Arms: CP-945,598
Drug: CP-945,598 Treatment B — Subjects receive CP-945,598 plus non-pharmacological weight loss program.
  Arms: CP-945,598 Treatment B

SUMMARY:
The purpose of this study is to determine if CP-945,598 is effective in the treatment of obesity in type 2 diabetic patients.

DETAILED DESCRIPTION:
The CP-945,598 program was terminated on November 3, 2008 due to changing regulatory perspectives on the risk/benefit profile of the CB1 class and likely new regulatory requirements for approval. No safety issues were involved in the termination decision.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be overweight (BMI 27- 50 kg/m2)
* Subjects must have type 2 diabetes mellitus

Exclusion Criteria:

* Pregnancy
* Serious or unstable current or past medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 975 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from baseline. | 1 year

SECONDARY OUTCOMES:
Proportion of subjects who lose 5 and 10% baseline body weight at 1 year; | 1 year
Proportion of subjects achieving HbA1c <6.5% and <7% at 1 year; | 1 year
Change from baseline in waist circumference at 1 year; | 1 year
Change from baseline fasting triglyceride and HDL concentrations at 1 year; | 1 year
Change from baseline in Total cholesterol, LDL, TNF α, adiponectin, and hsCRP levels at month 6 and 1 year; | 1 year
Change in prevalence of metabolic syndrome based on accepted definition at the time of study completion; | 1 year
HOMA IR (HOMA IR=fasting insulin x fasting glucose/22.5) at 1 year; | 1 year
Percentage of subjects who require additional diabetes pharmacotherapy because they meet protocol criteria for inadequate glycemic control; | 1 year
Population pharmacokinetic analysis of data acquired at trough and by randomized sparse sampling and exploration of PK/PD relationships; | 1 year
Change from baseline fasting plasma glucose concentration at 1 year; | 1 year
Change from baseline in Patient Health Questionnaire 9 and Generalized Anxiety Disorder 7 scores at months 1, 2, 3, 5, 6, 9, and 1 year; | 1 year
Change from baseline in background sulfonylurea or meglitinide dose requirements in subjects taking these medications; | 1 year
Change from baseline in 7 point home glucose profiles in a subset of subjects at 1 year; | 1 year
Primary and key secondary endpoints at any measured intermediate time points including weight at week 2, months 1, 6, 9, and 11; | 1 year
HbA1c, fasting plasma glucose at months 1, 3, 6, and 9; | 1 year
Waist circumference at months 3, 6, and 9; | 1 year
Fasting triglyceride and HDL concentrations at month 6 and patient reported outcome subscales: uncontrolled eating/hunger, power of food, physical functioning, and self esteem at months 3 and 6; | 1 year
Change from baseline in laboratory tests and ECGs at 1 year; vitals signs at (at Week 2, Months 1 - 6, 9, 11 and 1 year) and adverse events; | 1 year
Change in fasting and postprandial insulin concentrations determined from OGTT in a subset of subjects at 1 year; | 1 year
Protocol defined hypoglycemia event rates and proportion of subjects with hypoglycemic events; | 1 year
Change from baseline postprandial glucose determined from OGTT in a subset of subjects at 1 year; | 1 year
Changes from baseline in patient reported outcome subscales: uncontrolled eating/hunger, power of food, physical functioning, and self esteem at 1 year; | 1 year
Changes in patient reported outcome subscales not identified as key secondary endpoints at months 3, 6, and 12 | 1 year
Change from baseline HbA1c to 1 year; | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (83):
- United States (40):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Auburn, Maine
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bay City, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Morgantown, West Virginia
- Pfizer Investigational Site, Buenos Aires, Argentina
- Australia (5):
  - Pfizer Investigational Site, Garran, Australian Capital Territory
  - Pfizer Investigational Site, Wollongong, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Box Hill, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
- Brazil (3):
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (7):
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, L'Ancienne-Lorette, Quebec
  - Pfizer Investigational Site, Saint-Marc-des-Carrieres, Quebec
- Czechia (5):
  - Pfizer Investigational Site, Břeclav
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 4 - Krc
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Mittweida
- Mexico (4):
  - Pfizer Investigational Site, Tampico, Cd. Madero
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Slovakia (4):
  - Pfizer Investigational Site, Bratislava, Slovakia
  - Pfizer Investigational Site, Ľubochňa, Slovakia
  - Pfizer Investigational Site, Nitra, Slovakia
  - Pfizer Investigational Site, Banská Bystrica
- Sweden (2):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Huddinge
- United Kingdom (6):
  - Pfizer Investigational Site, Edinburgh, Lothian
  - Pfizer Investigational Site, Bath, Somerset
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Dumfries
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Luton

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351022&StudyName=A%201-Year%20Study%20On%20The%20Effects%20Of%20CP-945%2C598%20For%20The%20Treatment%20Of%20Obesity%20In%20Overweight%20Type%202%20Diabetic%20Patients